CLINICAL TRIAL: NCT01930721
Title: Comparison of Incision Angle of Mediolateral Episiotomy at 40 and 60 Degrees
Acronym: IAME
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, malka amen, resident, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: incision angle of mediolateral
Record Dates: First submitted 2012-06-16; First posted 2013-08-29 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Obstetric Labor Complications
MeSH Terms: conditions — Obstetric Labor Complications | interventions — Episiotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- incision angle of 60 degrees (Experimental): episiotomy incision angle will be defined as 60 degree as measured before cutting.
  Interventions: Procedure: episiotomy
- incision angle 40 degree episiotomy (Experimental): incision angle of episiotomy will be defined as 40 degree as measured before cutting.
  Interventions: Procedure: episiotomy

INTERVENTIONS:
Procedure: episiotomy — incision angle of episiotomy will be 60 degrees.
  Arms: incision angle 40 degree episiotomy
Procedure: episiotomy — incision angle of episiotomy will be 40 degree before cutting.
  Arms: incision angle of 60 degrees

SUMMARY:
The angle at which an episiotomy can be made is a continuous variable. If the investigators consider midline to be 0 degrees and a lateral episiotomy (never used today) to be 90 degrees, then it is theoretically possible to choose any angle from 0 to 90 degrees.

DETAILED DESCRIPTION:
Episiotomy is a surgical incision to the perineum in order to enlarge the vaginal orifice during the second stage of labor. Although seven types of episiotomy have been described in the literature , the most frequently performed types are the mediolateral and median episiotomies, with the former being the most common one. Despite being a common obstetric practice, the exact definition of a "mediolateral" episiotomy is often unclear. Several studies and reports, however, stated that a significant proportion of the so-claimed mediolateral episiotomy were not actually mediolateral. The current trial compares two angles of mediolateral episiotomy , regarding the risk of third- and fourth-degree perineal tearing, episiotomy-related pain and dyspareunia in primiparous women at a large tertiary maternity center, namely Ain Shams University Maternity Hospital, Cairo, Egypt.

ELIGIBILITY:
Inclusion Criteria:

1. Primigravida with singleton pregnancy presenting by vertex.
2. Gestational age > 37 weeks
3. No instrumental delivery.
4. No fetal distress or any emergency

Exclusion Criteria:

1. Women had an episiotomy because of fetal distress and for technical reasons (emergency or episiotomy incised prior to the fetal head crowning the perineum.
2. Inability to understand the informed consent.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 330 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-08 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
and fourth degree perineal tears. | intraoperative
  DESCRIBING THIRD AND FOURTH degree perieneal tears as regarding repair and post operative pain

CONTACTS AND LOCATIONS:
Overall Officials: ADEL SH SLAH EL-DIN, MD, Principal Investigator — LECTURER
Locations (1):
- Ain Shams Unversity Hospitals, Cairo, Egypt

REFERENCES:
- [Derived] El-Din AS, Kamal MM, Amin MA. Comparison between two incision angles of mediolateral episiotomy in primiparous women: a randomized controlled trial. J Obstet Gynaecol Res. 2014 Jul;40(7):1877-82. doi: 10.1111/jog.12432. PMID 25056465